CLINICAL TRIAL: NCT06697873
Title: Effects of Rhythmic Stabilization With and Without Closed Kinetic Chain Exercises on Upper Body Strength, Endurance and Balance Among Fast Bowlers
Brief Title: Effects of Rhythmic Stabilization With and Without Closed Kinetic Chain Exercises Among Fast Bowlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0402
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Sports Physical Therapy
Keywords: Balance; Rhythmical Exercise; Strength Training; Endurance; Physical

STUDY DESIGN:
Intervention Model Description: Assignment randomized control design
Who Masked: Participant
Masking Description: Double participant/investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group:A (Experimental): 21 participants will receive both Rhythmical stabilization and closed chain kinetic exercise followed by a warm up session with stretching 5 minutes and cool down session with 5 minutes
  Interventions: Other: Experimental Group: A
- Experimental Group:B (Experimental): 21 participants will receive Rhythmical stabilization training program followed by a warm up session with stretching 5 minutes and cool down session with 5 minutes.
  Interventions: Other: Experimental: Group B

INTERVENTIONS:
Other: Experimental Group: A — 21 participants will receive both Rhythmical stabilization and closed chain kinetic exercise followed by a warm up session with stretching 5 minutes and cool down session with 5 minutes
  Arms: Experimental Group:A
Other: Experimental: Group B — 21 participants will receive Rhythmical stabilization training program followed by a warm up session with stretching 5 minutes and cool down session with 5 minutes.
  Arms: Experimental Group:B

SUMMARY:
Effects of Rhythmic stabilization with and without Closed Kinetic Chain Exercises on upper body strength, endurance and balance among fast bowlers

DETAILED DESCRIPTION:
The literature mostly ignores the specific needs of fast bowlers in favor of concentrating on general strength and fitness for cricket players. Exercises for rhythmical stabilization, which improve neuromuscular control and stability, are not given much attention. There is not enough research done on closed chain workouts in cricket-specific contexts. Closed chain exercises replicate the weight transfer and ground response forces during quick bowling. There is a paucity of literature offering fast bowlers-specific evidence-based training routines, despite the unique demands of cricket. Coaches and practitioners are less able to create interventions that target the specifics of the fast bowling motion in the literature because there aren't many exercises specifically designed for cricket.

ELIGIBILITY:
Inclusion Criteria: Male athlete (16) Age of 18-35 years (17) Minimum of 6 months training experience (18) Healthy weight with BMI in category of 18.5 to 24.9 (15).

-

Exclusion Criteria: Joint or bone disease such as rheumatoid arthritis or osteoarthritis of the upper extremity (19).

Cervical spine pathology (20) Serious injury or history of surgery in the past year Any recent upper limb fracture Chronic limb discomfort or limitations that had a negative effect on exercises (e.g., shoulder pain and lateral epicondylitis) (20) Shoulder instability to be tested via load and shift test (21).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
1 repetition maximum bench press test (1RM) | 8 weeks
  The participant laid in a supine position with chin at the level of the padded surface of the bench. The starting position is when the hands are grasped slightly wider (~5cm) than the shoulder width and arms fully extended. From this position the weights pulled upwards with the elbows leading the barbell struck the underside of the bench and lowered to starting position. The posture to be adapted in bench press is as follows subject lays supine on the bench with eyes to be locked on the bar and the feet were planted on the ground with the lumbar region arched. The hand grip is to be 1.5 times the shoulder's width. The barbell is to be removed from the rack, lowered and to be paused briefly before being racked. A spotter is to be always placed behind the athlete
Repetitive push up test | 8 weeks
  The push up floor exercise is to be performed on a flat, stable surface, with the hands placed wider than the shoulder width. The body is aligned to the floor. For the repetition to be counted the athlete must go in a full range of motion, and the formation of 900 at the elbow at the end of the eccentric phase of the exercise
Closed Kinetic Chain Upper Extremity Stability Test (CKCUES Test) | 8 weeks
  CKCUEST is used for the evaluation of upper extremity strength, endurance and closed kinetic chain. The execution of the test is as follows. In push up position the two hands are to be placed at 90 cm, then one hand is to extend, and reach touch the other hands within a time of 15 seconds
Upper extremity Y-Balance Test | 8 weeks
  The YBT is a simple balance testing method to identify injury risks and functional asymmetries in an athlete. Each upper extremity is tested separately. The 3 lines each have a 1350 angle. The participant is placed in a push up position with the base of the proximal 3rd metacarpophalangeal joint placed at the center of the y balance board. The participant moves the hand in all 3 directions (medial, inferolateral and superolateral directions) as shown in the second figure below.

CONTACTS AND LOCATIONS:
Overall Officials: Ahad Hussain, DPT, Principal Investigator — Riphah Internation Univeersity
Locations (1):
- Pakistan Sports Academy, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catikkas F, Kurt C, Atalag O. Kinanthropometric attributes of young male combat sports athletes. Coll Antropol. 2013 Dec;37(4):1365-8. PMID 24611359
- [Background] da Silva BV, Simim MA, Marocolo M, Franchini E, da Mota GR. Optimal load for the peak power and maximal strength of the upper body in Brazilian Jiu-Jitsu athletes. J Strength Cond Res. 2015 Jun;29(6):1616-21. doi: 10.1519/JSC.0000000000000799. PMID 25486298
- [Background] Kizilay F, Cengiz DU. A comparison of functional vestibulo-ocular reflex and proprioception in athletes of combat sports and ball sports. Heliyon. 2023 Jun 25;9(7):e17540. doi: 10.1016/j.heliyon.2023.e17540. eCollection 2023 Jul. PMID 37455947
- [Background] Singla D, Hussain ME. Variations in cricket players' upper body dynamic balance across different levels of competition. Int J Adolesc Med Health. 2020 Jun 1;33(5). doi: 10.1515/ijamh-2019-0015. PMID 32474453
- [Background] Vaidya SS, Agarwal B, Singh Y, Mullerpatan R. Effect of Yoga on Performance and Physical Fitness in Cricket Bowlers. Int J Yoga Therap. 2021 Jan 1;31(1):Article_10. doi: 10.17761/2021-D-20-00060. PMID 34551075
- [Background] Herridge R, Turner A, Bishop C. Monitoring Changes in Power, Speed, Agility, and Endurance in Elite Cricketers During the Off-Season Period. J Strength Cond Res. 2020 Aug;34(8):2285-2293. doi: 10.1519/JSC.0000000000002077. PMID 28658073
- [Background] Doma K, Leicht A, Woods C, Harrison D, McGuckin T, Connor J. Effect of Exercise-Induced Muscle Damage on Bowling-Specific Motor Skills in Male Adolescent Cricketers. Sports (Basel). 2021 Jul 19;9(7):103. doi: 10.3390/sports9070103. PMID 34357937
- [Background] Ramachandran AK, Singh U, Connor JD, Doma K. Biomechanical and physical determinants of bowling speed in cricket: a novel approach to systematic review and meta-analysis of correlational data. Sports Biomech. 2024 Mar;23(3):347-369. doi: 10.1080/14763141.2020.1858152. Epub 2021 Jan 11. PMID 33428558
- [Background] Dionisio VC, de Baptista CRJA, Rodrigues AS, de Souza LAPS. Is it possible to stabilize the trunk using rhythmic stabilization in the upper limb? A cross-sectional study of asymptomatic individuals. J Man Manip Ther. 2018 Aug;26(4):212-217. doi: 10.1080/10669817.2018.1467994. Epub 2018 May 7. PMID 30083044
- [Background] Pozzi F, Plummer HA, Sanchez N, Lee Y, Michener LA. Electromyography activation of shoulder and trunk muscles is greater during closed chain compared to open chain exercises. J Electromyogr Kinesiol. 2022 Feb;62:102306. doi: 10.1016/j.jelekin.2019.05.007. Epub 2019 May 12. PMID 31151784
- See also: Kinanthropometric attributes of young male combat sports athletes. Collegium antropologicum. — https://pubmed.ncbi.nlm.nih.gov/24611359/